CLINICAL TRIAL: NCT02182284
Title: An Open-label, Randomized, Crossover Relative Bioavailability Study of a New Soft Gelatin Capsule Formulation of BI 201335 NA Compared to the Current Solution Formulation (Powder in Bottle (PIB), After Single Dose Oral Administration in Healthy Volunteers
Brief Title: Bioavailability of Soft Gelatin Capsule Formulation of BI 201335 NA Compared to the Solution Formulation in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1220.10
Record Dates: First submitted 2014-07-02; First posted 2014-07-08 (Estimated); Last update posted 2014-07-18 (Estimated); Status verified 2014-07

CONDITIONS: Healthy

ARMS (2):
- BI 201335 NA - low dose (Experimental)
  Interventions: Drug: low dose BI 201335 NA soft gelatine capsule (SGC); Drug: low dose BI 201335 NA powder in bottle (PIB)
- BI 201335 NA - high dose (Experimental)
  Interventions: Drug: high dose BI 201335 NA soft gelatine capsule (SGC); Drug: high dose BI 201335 NA powder in bottle (PIB)

INTERVENTIONS:
Drug: low dose BI 201335 NA soft gelatine capsule (SGC)
  Arms: BI 201335 NA - low dose
Drug: high dose BI 201335 NA soft gelatine capsule (SGC)
  Arms: BI 201335 NA - high dose
Drug: low dose BI 201335 NA powder in bottle (PIB)
  Arms: BI 201335 NA - low dose
Drug: high dose BI 201335 NA powder in bottle (PIB)
  Arms: BI 201335 NA - high dose

SUMMARY:
The objective of this study was to establish the relative bioavailability of a new soft gelatin capsule (SGC) formulation of BI 201335 NA compared to the current solution formulation (powder in bottle, PIB) for two doses (40 mg, 240 mg) in a parallel, two-way cross-over study design.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females according to the following criteria: Based upon a complete medical history, including the physical examination, vital signs (blood pressure (BP), pulse rate (PR)), 12-lead ECG (electrocardiogram), clinical laboratory tests
* Age ≥18 and Age ≤50 years
* Body Mass Index (BMI) ≥18.5 and BMI ≤29.9 kg/m2
* Signed and dated written informed consent prior to admission to the study in accordance with GCP (Good Clinical Practice) and the local legislation

Exclusion Criteria:

* Any finding from the medical examination (including BP, PR and ECG) deviating from normal and of clinical relevance, as assessed by the investigator
* Any evidence of a clinically relevant concomitant disease
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Surgery of the gastrointestinal tract (except appendectomy)
* Chronic or relevant acute infections
* History of relevant allergy/hypersensitivity (including allergy to drug or its excipients)
* Concomitant drugs that in the opinion of the investigator (in consultation with the BI medical monitor or pharmacokinetics), would have interfered with the adsorption, distribution or metabolism of BI 201335
* Use of drugs which might reasonably influence the results of the trial or that prolong the QT/QTc (corrected QT interval) interval within 30 days prior to screening until trial completion
* Use of any investigational drug within 30 days prior to enrolment; or the planned usage of any investigational drug during the course of the current study
* Smoking (>10 cigarettes or >3 cigars or >3 pipes/day)
* Inability to abstain from alcohol from Day -14 to day 22
* Drug abuse
* Blood donation (more than 100 mL within four weeks prior to administration or during the trial)
* Excessive physical activities (within one week prior to administration or during the trial)
* Any laboratory value outside the reference range that is of clinical relevance at screening, according to the judgement of the investigator
* A marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval >450 ms)
* Infected with hepatitis A, hepatitis B or hepatitis C viruses (defined as either being hepatitis A antibody positive, hepatitis B surface antigen or HBV DNA positive, or hepatitis C antibody positive)
* Positive ELISA for HIV-1 (Human immunodeficiency virus) or HIV-2
* For female subjects:

  * Pregnancy or planning to become pregnant within 2 months of study completion
  * Positive pregnancy test
  * No adequate contraception, e.g. sterilisation, IUD (intrauterine device), have not been using a barrier method of contraception for at least 3 months prior to participation in the study
  * Are not willing or are unable to use a reliable method of barrier contraception (such as diaphragm with spermicidal cream/jelly or condoms with spermicidal foam), during and up to 2 months after completion/termination of the trial
  * Lactation period

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2008-01; Primary Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
AUC0-∞ (area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) | Before and 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 16, 24, 36, 48, 72, 96, 120 hours after administration of study drug
Cmax (measured maximum concentration of the analyte in plasma) | Before and 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 16, 24, 36, 48, 72, 96, 120 hours after administration of study drug

SECONDARY OUTCOMES:
tmax (time from dosing to the maximum concentration of the analyte in plasma) | Before and 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 16, 24, 36, 48, 72, 96, 120 hours after administration of study drug
AUC0-tz (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the time of the last quantifiable data point) | Before and 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 16, 24, 36, 48, 72, 96, 120 hours after administration of study drug
t1/2 (terminal half-life of the analyte in plasma) | Before and 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 16, 24, 36, 48, 72, 96, 120 hours after administration of study drug
CL/F (apparent clearance of the analyte in the plasma after oral administration) | Before and 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 16, 24, 36, 48, 72, 96, 120 hours after administration of study drug
λz (terminal elimination rate constant in plasma) | Before and 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 16, 24, 36, 48, 72, 96, 120 hours after administration of study drug
MRTpo (mean residence time of the analyte in the body after oral administration) | Before and 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 16, 24, 36, 48, 72, 96, 120 hours after administration of study drug
Vz/F (apparent volume of distribution during the terminal phase λz following an oral dose) | Before and 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 16, 24, 36, 48, 72, 96, 120 hours after administration of study drug
C24 (measured concentration of the analyte in plasma 24 hours after oral administration) | Before and 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 16, 24, 36, 48, 72, 96, 120 hours after administration of study drug
Number of patients with clinically significant changes in vital signs | Baseline, days 1-6 of each treatment period and day 22
Number of patients with abnormal changes in laboratory parameters | Baseline, days 1 and 3-6 of each treatment period and day 22
Number of patients with adverse events | up to 29 days